CLINICAL TRIAL: NCT02443506
Title: A Randomized Double-blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 623 Following Single Dose Administration in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study to Examine the Safety, Pharmacokinetics and Pharmacodynamics of Single Dose of AMG 623 in Subjects With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20040147
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-04

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 623 (Experimental): Single dose of AMG 623 administered as subcutaneous and intravenous doses
  Interventions: Drug: AMG 623
- Placebo (Placebo Comparator): Single dose of matching AMG 623 placebo administered as subcutaneous and intravenous doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 623 — Single dose of AMG 623 administered as subcutaneous and intravenous doses
  Arms: AMG 623
Drug: Placebo — Single dose of matching AMG 623 placebo administered as subcutaneous and intravenous doses
  Arms: Placebo

SUMMARY:
This study is to evaluate the safety of AMG 623 in subjects with systemic lupus erythematosus. The study consists of a 21 day screening period followed by administration of the investigational product and up to 70 day follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between the ages of 18 and 55
* Diagnosis of SLE
* Have had a disease duration of at least 1 year, as diagnosed by a physician

Exclusion Criteria:

* Have a disorder (including psychiatric), condition or clinically significant disease (other than a diagnosis of SLE) that would interfere with the study evaluation, completion and/or procedures per the investigator's discretion
* Have active vasculitis, active CNS lupus requiring therapy, active acute renal disease, uncontrolled hypertension, uncontrolled diabetes or active systemic infection
* Have had signs or symptoms of viral or bacterial infection within 30 days of enrollment
* Have received a daily dose of greater than 10 mg prednisone (or equivalent) in the prior 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2004-10; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | up to 70 days
Incidence of abnormal clinically significant vital signs | up to 70 days
Incidence of abnormal clinically significant chemistry, hematology and urinalysis test results | up to 70 days
Incidence of abnormal clinically significant ECG results | up to 70 days

SECONDARY OUTCOMES:
Pharmacokinetics profile of AMG 623 including Tmax, AUClast and Cmax | up to 70 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Stohl W, Merrill JT, Looney RJ, Buyon J, Wallace DJ, Weisman MH, Ginzler EM, Cooke B, Holloway D, Kaliyaperumal A, Kuchimanchi KR, Cheah TC, Rasmussen E, Ferbas J, Belouski SS, Tsuji W, Zack DJ. Treatment of systemic lupus erythematosus patients with the BAFF antagonist "peptibody" blisibimod (AMG 623/A-623): results from randomized, double-blind phase 1a and phase 1b trials. Arthritis Res Ther. 2015 Aug 20;17(1):215. doi: 10.1186/s13075-015-0741-z. PMID 26290435
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com